CLINICAL TRIAL: NCT03329001
Title: An Open-Label, Randomized-Sequence, Multicenter, Single-Crossover Study to Assess the Relative Bioavailability and Bioequivalence of Niraparib Tablet Formulation Compared to Niraparib Capsule Formulation in Patients With Advanced Solid Tumors
Brief Title: Crossover Study to Assess the Relative Bioavailability and Bioequivalence of Niraparib Tablet Compared to Niraparib Capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 213362; 3000-01-004 (Other: Tesaro)
Record Dates: First submitted 2017-10-23; First posted 2017-11-01 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Neoplasms
Keywords: PARP inhibitor; niraparib; Solid Tumor; Zejula
MeSH Terms: conditions — Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Stage 1: Tablet-Capsule Sequence (Experimental): Single dose niraparib tablet followed by single dose niraparib capsule followed by optional daily dosing extension phase
  Interventions: Drug: Niraparib Tablet; Drug: Niraparib Capsule
- Stage 1: Capsule-Tablet Sequence (Experimental): Single dose niraparib capsule followed by single dose niraparib tablet followed by optional daily dosing extension phase
  Interventions: Drug: Niraparib Tablet; Drug: Niraparib Capsule
- Stage 2: Tablet-Capsule Sequence (Experimental): Single dose niraparib tablet followed by single dose niraparib capsule followed by optional daily dosing extension phase.
  Interventions: Drug: Niraparib Tablet; Drug: Niraparib Capsule
- Stage 2: Capsule-Tablet Sequence (Experimental): Single dose niraparib capsule followed by single dose niraparib tablet followed by optional daily dosing extension phase
  Interventions: Drug: Niraparib Tablet; Drug: Niraparib Capsule
- Stage 3: High fat meal-fasted sequence (Experimental): Single dose niraparib tablet with a high fat meal followed by single dose of niraparib tablet in a fasted state.
  Interventions: Drug: Niraparib Tablet
- Stage 3: Fasted-high fat meal sequence (Experimental): Single dose niraparib tablet in a fasted state followed by single dose Niraparib tablet with a high fat meal.
  Interventions: Drug: Niraparib Tablet

INTERVENTIONS:
Drug: Niraparib Tablet — Niraparib tablet formulation
Drug: Niraparib Capsule — Niraparib capsule formulation
  Arms: Stage 1: Capsule-Tablet Sequence; Stage 1: Tablet-Capsule Sequence; Stage 2: Capsule-Tablet Sequence; Stage 2: Tablet-Capsule Sequence

SUMMARY:
This is a three stage, open label, randomized-sequence, single-crossover Phase 1 study to evaluate the relative bioavailability (BA) and Bioequivalence (BE) of niraparib administered as a tablet formulation compared to the reference capsule formulation currently marketed in the United States. Stage 3 evaluates the effect of a high-fat meal on niraparib pharmacokinetics (PK) following a single dose of the tablet. The Extension Phase of this study is to enable participants enrolled in the study to continue to receive treatment with niraparib tablets if they are tolerating it and, in the Investigator's opinion, may receive benefit.

ELIGIBILITY:
Key inclusion criteria:

PK Phase: To be considered eligible to participate in this study, all of the following requirements must be met:

* Participants with histologically or cytologically confirmed diagnosis of metastatic or locally advanced solid tumors that have failed to respond to standard therapy, has progressed despite standard therapy, or for which no standard therapy exists, and who may benefit from treatment with a poly (adenosine diphosphate-ribose) polymerase (PARP) inhibitor as assessed by the Investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Adequate organ function as defined: Absolute neutrophil count ≥ 1,500 per microliter (/μL) (For Stage 3: >=1000/μL); Platelets ≥ 100,000/μL; Hemoglobin ≥ 9 grams per deciliter (g/dL) (5.6 millimolar [mM]); Serum creatinine ≤ 1.5 × the upper limit of normal (ULN) or a calculated creatinine clearance ≥ 60 milliliters per minute (mL/min) using the Cockcroft-Gault equation or 24-hour urine creatinine clearance.; Total bilirubin ≤ 1.5 × ULN except in participants with Gilbert's syndrome. Participants with Gilbert's syndrome may enroll if direct bilirubin ≤ 1.5 × ULN of the direct bilirubin; Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN unless liver metastases are present, in which case, they must be ≤ 5 × ULN.
* Participant has recovered to Grade 1 toxicity from prior cancer therapy (a participant with Grade 2 neuropathy or Grade 2 alopecia is an exception to this criterion and may qualify for this study).
* Female participant of childbearing potential is not breastfeeding, has a negative serum pregnancy test within 72 hours prior to taking study drug and agrees to abstain from activities that could result in pregnancy from Screening through 180 days after the last dose of study drug.
* Male participant agrees to use an adequate method of contraception and not donate sperm starting with the first dose of study drug through 90 days after the last dose of study drug.
* (For Stage 3): CNS inclusion - Based on screening brain magnetic resonance imaging indicating no evidence of brain metastasis or needing immediate local therapy.
* Participant is able to eat a high fat meal.
* Participant is able to fast for a minimum of 10 hours before start of visit and for an additional 4 hours after study visit.

Extension Phase:

* ECOG performance status of 0 to 2.
* Adequate organ function as defined: Absolute neutrophil count ≥ 1,500/μL (For Stage 3: >=1000/μL); Platelets ≥ 100,000/μL; Hemoglobin ≥ 9 g/dL (5.6 mM); serum creatinine ≤ 1.5 × the ULN or a calculated creatinine clearance ≥ 60 mL/min (For Stage 3: ≥ 30 mL/min) using the Cockcroft-Gault equation or 24-hour urine creatinine clearance; Total bilirubin ≤ 1.5 × ULN except in participant with Gilbert's syndrome. Participants with Gilbert's syndrome may enroll if direct bilirubin ≤ 1.5 × ULN of the direct bilirubin; AST and ALT ≤ 2.5 × ULN unless liver metastases are present, in which case, they must be ≤5 × ULN
* Female participant of childbearing potential is not breastfeeding, has a negative serum pregnancy test within 72 hours prior to taking study drug and agrees to abstain from activities that could result in pregnancy from Screening through 180 days after the last dose of study drug.
* Male participant agrees to use an adequate method of contraception and not donate sperm starting with the first dose of study drug through 90 days after the last dose of study drug.

Key Exclusion Criteria: PK Phase:

* Known diagnosis of immunodeficiency
* Symptomatic uncontrolled brain or leptomeningeal metastases.
* Major surgery within 3 weeks of starting the study or participant has not recovered from any effects of any major surgery.
* Participant is considered a poor medical risk due to a serious, uncontrolled medical disorder; nonmalignant systemic disease; or active, uncontrolled infection.
* Known history of myelodysplastic syndrome or acute myeloid leukemia.
* Participant is currently taking any of the following P-glycoprotein (P-gp) inhibitors: amiodarone, azithromycin, captopril, carvedilol, clarithromycin, conivaptan, cyclosporine, diltiazem, dronedarone, erythromycin, felodipine, itraconazole, ketoconazole, lopinavir and ritonavir, quercetin, quinidine, ranolazine, ticagrelor, and verapamil (Does not apply for Extension Phase).
* Participant taking proton pump inhibitors, antacids, or histamine 2 blockers within 48 hours prior to study drug administration (Does not apply for Extension Phase).
* Participant has gastric, gastro-esophageal or esophageal cancer; participant is unable to swallow orally administered medication; or participant has gastrointestinal disorders or significant gastrointestinal resection likely to interfere with the absorption of niraparib.
* Participant has known active hepatic disease
* Participant has a past or current history of chronic alcohol use.
* Participant has significant pleural effusion or ascites that is expected to require drainage during the PK Phase (Does not apply for Extension Phase).
* For Stage 3 only: Participant is currently taking a lipase inhibitor or cholesterol absorption inhibitor, such as orlistat or ezetimibe, respectively. (Does not apply for participation in Extension Phase of this study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- United States (16):
  - GSK Investigational Site, Encinitas, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, San Marcos, Texas

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data (IPD) and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Background] Falchook G, Patnaik A, Richardson DL, Harvey RD, Sharma MR, Hafez N, Hamilton E, Piha-Paul SA, Barve M, Wise-Draper T, Patel MR, Dowlati A, Pascuzzo J, Tang SC, Faltermeier C, Malinowska IA, Shtessel L, Striha A, Potocka E. A Relative Bioavailability, Bioequivalence, and Food Effect Study of Niraparib Tablets in Patients with Advanced Solid Tumors. Clin Ther. 2024 Mar;46(3):228-238. doi: 10.1016/j.clinthera.2024.01.004. Epub 2024 Feb 28. PMID 38423866

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 3-stage, single cross-over study. The study had a pharmacokinetic (PK) phase consisting of stages 1, 2, and 3 and an Extension Phase. The Extension Phase based on Investigator and Sponsor's decision provided qualifying participants continued access to niraparib therapy.
Pre-assignment Details: A total of 236 participants were enrolled. The Safety Population comprised all participants who received any amount of niraparib during the PK Phase and Extension Phase of the study.
Groups:
- Stage 1: Niraparib Tablet/Capsule: Participants received a single oral dose of 300 milligrams (mg) niraparib tablet in a fasted state in Period 1, followed by a wash-out period of 7 days. In Period 2, participants received a single oral dose of 3 capsules of 100 mg niraparib in a fasted state followed by a 7-day wash-out period. After the last dose of niraparib, participants who did not enter the Extension Phase were followed for up to 30 days (safety follow-up [f/u]) while participants eligible for Extension Phase proceeded for Extension Phase screening. Eligible participants then entered the Extension Phase, where they received 300 mg or 200 mg niraparib tablets or capsules for once daily dosing depending on their body weight and platelet count.
- Stage 1: Niraparib Capsule/Tablet: Participants received a single oral dose of 3x100 mg niraparib capsules in a fasted state in Period 1, followed by a wash-out period of 7 days. In Period 2, participants received a single oral dose of 300 mg niraparib tablet in a fasted state followed by a 7-day wash-out period. After the last dose of niraparib, participants who did not enter the Extension Phase were followed for up to 30 days (safety f/u) while participants eligible for Extension Phase proceeded for Extension Phase screening. Eligible participants then entered the Extension Phase, where they received 300 mg or 200 mg niraparib tablets or capsules for once daily dosing depending on their body weight and platelet count.
- Stage 2: Niraparib Tablet/Capsule: Participants received a single oral dose of 300 mg niraparib tablet in a fasted state in Period 1, followed by a wash-out period of 14 days. In Period 2, participants received a single oral dose of 3 capsules of 100 mg niraparib in a fasted state followed by a 7-day wash-out period. After the last dose of niraparib, participants who did not enter the Extension Phase were followed for up to 30 days (safety f/u) while participants eligible for Extension Phase proceeded for Extension Phase screening. Eligible participants then entered the Extension Phase, where they received 300 mg or 200 mg niraparib tablets or capsules for once daily dosing depending on their body weight and platelet count.
- Stage 2: Niraparib Capsule/Tablet: Participants received a single oral dose of three 100 mg niraparib capsules in a fasted state in Period 1, followed by a wash-out period of 14 days. In Period 2, participants received a single oral dose of 300 mg niraparib tablet in a fasted state followed by a 7-day wash-out period. After the last dose of niraparib, participants who did not enter the Extension Phase were followed for up to 30 days (safety f/u) while participants eligible for Extension Phase proceeded for Extension Phase screening. Eligible participants then entered the Extension Phase, where they received 300 mg or 200 mg niraparib tablets or capsules for once daily dosing depending on their body weight and platelet count.
- Stage 3: Niraparib Tablet Fasted/Fed: Participants received a single oral dose of 300 mg niraparib tablet in a fasted state in Period 1, followed by a wash-out period of 14 days. In period 2, participants received a single oral dose of 300 mg niraparib tablet in a fed state with a high fat meal followed by a 7-day wash-out period. After the last dose of niraparib, participants who did not enter the Extension Phase were followed for up to 30 days (safety f/u) while participants eligible for Extension Phase proceeded for Extension Phase screening. Eligible participants then entered the Extension Phase, where they received 300 mg or 200 mg niraparib tablets or capsules for once daily dosing depending on their body weight and platelet count.
- Stage 3: Niraparib Tablet Fed/Fasted: Participants received a single oral dose of 300 mg niraparib tablet in a fed state with a high fat meal in Period 1, followed by a wash-out period of 14 days. In period 2, participants received a single oral dose of 300 mg niraparib tablet in a fasted state followed by a 7-day wash-out period. After the last dose of niraparib, participants who did not enter the Extension Phase were followed for up to 30 days (safety f/u) while participants eligible for Extension Phase proceeded for Extension Phase screening. Eligible participants then entered the Extension Phase, where they received 300 mg or 200 mg niraparib tablets or capsules for once daily dosing depending on their body weight and platelet count.
- Extension Phase: Niraparib Tablet: Participants received starting dose of 300 mg or 200 mg of niraparib tablet for QD dosing orally or 3 x 100 mg or 2 x 100 mg for QD niraparib tablets dosing orally in the Extension Phase based on participant's baseline actual body weight or platelet count.
- Extension Phase: Niraparib Capsule: Participants received starting dose of 300 mg or 200 mg of niraparib capsules for QD dosing orally or 3 x 100 mg or 2 x 100 mg for QD niraparib capsules dosing orally in the Extension Phase based on participant's baseline actual body weight or platelet count.
Period: Stage 1: PK Phase- Period 1 (Day 1)
Arm/Group | Stage 1: Niraparib Tablet/Capsule | Stage 1: Niraparib Capsule/Tablet | Stage 2: Niraparib Tablet/Capsule | Stage 2: Niraparib Capsule/Tablet | Stage 3: Niraparib Tablet Fasted/Fed | Stage 3: Niraparib Tablet Fed/Fasted | Extension Phase: Niraparib Tablet | Extension Phase: Niraparib Capsule
Started | 15 | 14 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 15 | 14 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage1:PK Phase Washout1(W)(Up to Day 7)
Arm/Group | Stage 1: Niraparib Tablet/Capsule | Stage 1: Niraparib Capsule/Tablet | Stage 2: Niraparib Tablet/Capsule | Stage 2: Niraparib Capsule/Tablet | Stage 3: Niraparib Tablet Fasted/Fed | Stage 3: Niraparib Tablet Fed/Fasted | Extension Phase: Niraparib Tablet | Extension Phase: Niraparib Capsule
Started | 15 | 14 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 15 | 14 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 1: PK Phase- Period 2 (Day 1)
Arm/Group | Stage 1: Niraparib Tablet/Capsule | Stage 1: Niraparib Capsule/Tablet | Stage 2: Niraparib Tablet/Capsule | Stage 2: Niraparib Capsule/Tablet | Stage 3: Niraparib Tablet Fasted/Fed | Stage 3: Niraparib Tablet Fed/Fasted | Extension Phase: Niraparib Tablet | Extension Phase: Niraparib Capsule
Started | 15 | 14 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 15 | 14 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage1:PK Phase W2 (Up to Day 7)
Arm/Group | Stage 1: Niraparib Tablet/Capsule | Stage 1: Niraparib Capsule/Tablet | Stage 2: Niraparib Tablet/Capsule | Stage 2: Niraparib Capsule/Tablet | Stage 3: Niraparib Tablet Fasted/Fed | Stage 3: Niraparib Tablet Fed/Fasted | Extension Phase: Niraparib Tablet | Extension Phase: Niraparib Capsule
Started | 15 | 14 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 15 | 14 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 2: PK Phase-Period 1 (Day 1)
Arm/Group | Stage 1: Niraparib Tablet/Capsule | Stage 1: Niraparib Capsule/Tablet | Stage 2: Niraparib Tablet/Capsule | Stage 2: Niraparib Capsule/Tablet | Stage 3: Niraparib Tablet Fasted/Fed | Stage 3: Niraparib Tablet Fed/Fasted | Extension Phase: Niraparib Tablet | Extension Phase: Niraparib Capsule
Started | 0 | 0 | 90 | 89 | 0 | 0 | 0 | 0
Treatment Received | 0 | 0 | 85 | 83 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 85 | 83 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 5 | 6 | 0 | 0 | 0 | 0
Not completed — Randomized, but did not receive treatment | 0 | 0 | 5 | 6 | 0 | 0 | 0 | 0
Period: Stage 2: PK Phase-W1 (Up to Day 14)
Arm/Group | Stage 1: Niraparib Tablet/Capsule | Stage 1: Niraparib Capsule/Tablet | Stage 2: Niraparib Tablet/Capsule | Stage 2: Niraparib Capsule/Tablet | Stage 3: Niraparib Tablet Fasted/Fed | Stage 3: Niraparib Tablet Fed/Fasted | Extension Phase: Niraparib Tablet | Extension Phase: Niraparib Capsule
Started | 0 | 0 | 85 | 83 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 69 | 71 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 16 | 12 | 0 | 0 | 0 | 0
Not completed — Deemed unevaluable | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Sponsor discontinued the participant | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Sponsor and Investigator decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Participant had incorrectly overdosed and removed from PK phase | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Participant admitted to emergency room for elevated serum creatinine | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Participant unable to complete due to Tornado in site area | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Participant non-compliance | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Vomiting within protocol-specified hours of dose administration | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Disease progression per Investigator Decision | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 5 | 2 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Period: Stage 2: PK Phase- Period 2 (Day 15)
Arm/Group | Stage 1: Niraparib Tablet/Capsule | Stage 1: Niraparib Capsule/Tablet | Stage 2: Niraparib Tablet/Capsule | Stage 2: Niraparib Capsule/Tablet | Stage 3: Niraparib Tablet Fasted/Fed | Stage 3: Niraparib Tablet Fed/Fasted | Extension Phase: Niraparib Tablet | Extension Phase: Niraparib Capsule
Started | 0 | 0 | 69 | 71 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 69 | 71 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage2:PK Phase W2 (Up to Day 7)
Arm/Group | Stage 1: Niraparib Tablet/Capsule | Stage 1: Niraparib Capsule/Tablet | Stage 2: Niraparib Tablet/Capsule | Stage 2: Niraparib Capsule/Tablet | Stage 3: Niraparib Tablet Fasted/Fed | Stage 3: Niraparib Tablet Fed/Fasted | Extension Phase: Niraparib Tablet | Extension Phase: Niraparib Capsule
Started | 0 | 0 | 69 | 71 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 64 | 66 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 5 | 5 | 0 | 0 | 0 | 0
Not completed — Participant had paracentesis | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Participant forgot appointment | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Participant missed PK sampling in Period 1 Day 8 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Deemed unevaluable | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Participant was not in fasted state and therefore was outside of protocol compliance | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Disease progression per Investigator Decision | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Period: Stage 3: PK Phase- Period 1 (Day 1)
Arm/Group | Stage 1: Niraparib Tablet/Capsule | Stage 1: Niraparib Capsule/Tablet | Stage 2: Niraparib Tablet/Capsule | Stage 2: Niraparib Capsule/Tablet | Stage 3: Niraparib Tablet Fasted/Fed | Stage 3: Niraparib Tablet Fed/Fasted | Extension Phase: Niraparib Tablet | Extension Phase: Niraparib Capsule
Started | 0 | 0 | 0 | 0 | 14 | 14 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 11 | 12 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Clinical progression | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Stage 3: PK Phase-W1 (Up to Day 14)
Arm/Group | Stage 1: Niraparib Tablet/Capsule | Stage 1: Niraparib Capsule/Tablet | Stage 2: Niraparib Tablet/Capsule | Stage 2: Niraparib Capsule/Tablet | Stage 3: Niraparib Tablet Fasted/Fed | Stage 3: Niraparib Tablet Fed/Fasted | Extension Phase: Niraparib Tablet | Extension Phase: Niraparib Capsule
Started | 0 | 0 | 0 | 0 | 11 | 12 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 11 | 12 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 3: PK Phase- Period 2 (Day 15)
Arm/Group | Stage 1: Niraparib Tablet/Capsule | Stage 1: Niraparib Capsule/Tablet | Stage 2: Niraparib Tablet/Capsule | Stage 2: Niraparib Capsule/Tablet | Stage 3: Niraparib Tablet Fasted/Fed | Stage 3: Niraparib Tablet Fed/Fasted | Extension Phase: Niraparib Tablet | Extension Phase: Niraparib Capsule
Started | 0 | 0 | 0 | 0 | 11 | 12 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 10 | 11 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Vomiting within protocol-specified hours of dose administration | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Period: Stage3:PK Phase W2 (Up to Day 7)
Arm/Group | Stage 1: Niraparib Tablet/Capsule | Stage 1: Niraparib Capsule/Tablet | Stage 2: Niraparib Tablet/Capsule | Stage 2: Niraparib Capsule/Tablet | Stage 3: Niraparib Tablet Fasted/Fed | Stage 3: Niraparib Tablet Fed/Fasted | Extension Phase: Niraparib Tablet | Extension Phase: Niraparib Capsule
Started | 0 | 0 | 0 | 0 | 10 | 11 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 10 | 11 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Extension Phase(Approx 5 Years 5 Months)
Arm/Group | Stage 1: Niraparib Tablet/Capsule | Stage 1: Niraparib Capsule/Tablet | Stage 2: Niraparib Tablet/Capsule | Stage 2: Niraparib Capsule/Tablet | Stage 3: Niraparib Tablet Fasted/Fed | Stage 3: Niraparib Tablet Fed/Fasted | Extension Phase: Niraparib Tablet | Extension Phase: Niraparib Capsule
Started | 0 | 0 | 0 | 0 | 0 | 0 | 124 | 66
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 53 | 36
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 71 | 30
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 22 | 14
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 3
Not completed — Other reasons | 0 | 0 | 0 | 0 | 0 | 0 | 30 | 13

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were presented for Safety Population, all participants who received any amount of niraparib during the PK phase of study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1: Niraparib Tablet/Capsule | Stage 1: Niraparib Capsule/Tablet | Stage 2: Niraparib Tablet/Capsule | Stage 2: Niraparib Capsule/Tablet | Stage 3: Niraparib Tablet Fasted/Fed | Stage 3: Niraparib Tablet Fed/Fasted | Total
Number analyzed (Participants) | 15 | 14 | 85 | 83 | 14 | 14 | 225
Age, Customized [Count of Participants; unit: Participants]
  <18 to <65 years | 5 | 7 | 43 | 38 | 6 | 9 | 108
  >=65 to <75 years | 9 | 4 | 27 | 32 | 7 | 1 | 80
  >=75 years | 1 | 3 | 15 | 13 | 1 | 4 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 48 | 48 | 5 | 6 | 125
  Male | 6 | 5 | 37 | 35 | 9 | 8 | 100
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | 14 | 63 | 62 | 8 | 10 | 171
  African American | 1 | 0 | 11 | 11 | 5 | 0 | 28
  Asian | 0 | 0 | 5 | 3 | 0 | 0 | 8
  American Indian or Alaska Native | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Unknown | 0 | 0 | 4 | 7 | 1 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC[0-t]) for Niraparib-Stage 1 PK Phase
Description: Blood samples were collected at indicated time points for pharmacokinetic assessment of AUC(0-t). Pharmacokinetic parameters were calculated using standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose in each treatment period
Population: Bioavailability (BA) Evaluable Population included all participants who completed both PK Periods and had sufficient PK sample collection to accurately estimate PK parameters, without significant niraparib carryover (Baseline concentration >5 percent (%) of maximum observed plasma concentration [Cmax]), in both Periods.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Groups:
- Stage 1: Niraparib Tablet: Participants received a single oral dose of 300 mg niraparib tablet in a fasted state in either Period 1 or Period 2 of Stage 1 PK Phase.
- Stage 1: Niraparib Capsule: Participants received a single oral dose of 300 mg (3x100 mg capsules) niraparib in a fasted state in either Period 1 or Period 2 of Stage 1 PK Phase.
Arm/Group | Stage 1: Niraparib Tablet | Stage 1: Niraparib Capsule
Number analyzed (Participants) | 23 | 23
Hours*nanogram per milliliter | 14900 (43.0) | 16100 (41.3)
Statistical Analysis 1: Comparison: Stage 1: Niraparib Tablet vs Stage 1: Niraparib Capsule; Test type: Other; Ratio of geometric least square mean = 0.9110, 90% CI 2-sided [0.8550 to 0.9706] — Relative bioavailability (AUC[tablet]/AUC[capsule]) was assessed using analysis of variance (ANOVA) model accounting for sequence, participants nested with sequences, period and treatment

2. Primary Outcome: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC[0 to Inf]) for Niraparib-Stage 1 PK Phase
Description: Blood samples were collected at indicated time points for pharmacokinetic assessment of AUC(0 to inf). Pharmacokinetic parameters were calculated using standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose in each treatment period
Population: BA Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Stage 1: Niraparib Tablet | Stage 1: Niraparib Capsule
Number analyzed (Participants) | 23 | 23
Hours*nanogram per milliliter | 16200 (44.5) | 17200 (41.8)
Statistical Analysis 1: Comparison: Stage 1: Niraparib Tablet vs Stage 1: Niraparib Capsule; Test type: Other; Ratio of geometric least square mean = 0.9216, 90% CI 2-sided [0.8631 to 0.9841] — Relative bioavailability (AUC[tablet]/AUC[capsule]) was assessed using ANOVA model accounting for sequence, participants nested with sequences, period and treatment

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for Niraparib-Stage 1 PK Phase
Description: Blood samples were collected at indicated time points for pharmacokinetic assessment of Cmax. Pharmacokinetic parameters were calculated using standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose in each treatment period
Population: BA Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Stage 1: Niraparib Tablet | Stage 1: Niraparib Capsule
Number analyzed (Participants) | 23 | 23
Nanograms per milliliter | 451 (47.8) | 467 (50.0)
Statistical Analysis 1: Comparison: Stage 1: Niraparib Tablet vs Stage 1: Niraparib Capsule; Test type: Other; Ratio of geometric least square mean = 0.9483, 90% CI 2-sided [0.8489 to 1.0593] — Relative bioavailability (Cmax[tablet]/Cmax[capsule]) was assessed using ANOVA model accounting for sequence, participants nested with sequences, period and treatment

4. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for Niraparib-Stage 1 PK Phase
Description: Blood samples were collected at indicated time points for pharmacokinetic assessment of Tmax. Pharmacokinetic parameters were calculated using standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose in each treatment period
Population: BA Evaluable Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Stage 1: Niraparib Tablet | Stage 1: Niraparib Capsule
Number analyzed (Participants) | 23 | 23
Hours | 4.05 [1.98 to 8.00] | 4.00 [1.52 to 25.02]

5. Primary Outcome: Terminal Half-life (T1/2) for Niraparib-Stage 1 PK Phase
Description: Blood samples were collected at indicated time points for pharmacokinetic assessment of T1/2. Pharmacokinetic parameters were calculated using standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose in each treatment period
Population: BA Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Stage 1: Niraparib Tablet | Stage 1: Niraparib Capsule
Number analyzed (Participants) | 23 | 23
Hours | 47.3 (22.2) | 43.8 (23.1)

6. Primary Outcome: Apparent Total Body Clearance (CL/F) for Niraparib-Stage 1 PK Phase
Description: Blood samples were collected at indicated time points for pharmacokinetic assessment of CL/F. Pharmacokinetic parameters were calculated using standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose in each treatment period
Population: BA Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Stage 1: Niraparib Tablet | Stage 1: Niraparib Capsule
Number analyzed (Participants) | 23 | 23
Liters per hour | 18.5 (44.5) | 17.4 (41.8)

7. Primary Outcome: Apparent Terminal Volume of Distribution (Vz/F) for Niraparib-Stage 1 PK Phase
Description: Blood samples were collected at indicated time points for pharmacokinetic assessment of Vz/F. Pharmacokinetic parameters were calculated using standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose in each treatment period
Population: BA Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Stage 1: Niraparib Tablet | Stage 1: Niraparib Capsule
Number analyzed (Participants) | 23 | 23
Liters | 1260 (45.4) | 1100 (43.1)

8. Primary Outcome: AUC(0-t) for Niraparib-Stage 2 PK Phase
Description: as for outcome 1
Time Frame: Pre-dose, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose in each treatment period
Population: Bioequivalence (BE) Evaluable Population included all participants who completed both the Study Drug and Washout/PK and had sufficient PK sample collection to accurately estimate PK parameters, without significant niraparib carryover and without events or protocol deviations deemed affect PK, in both Periods. Only those participants with estimable PK parameter data in both periods were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Groups:
- Stage 2: Niraparib Tablet: Participants received a single oral dose of 300 mg niraparib tablet in a fasted state in either Period 1 or Period 2 of Stage 2 PK Phase.
- Stage 2: Niraparib Capsule: Participants received a single oral dose of 300 mg (3x100 mg capsules) niraparib in a fasted state in either Period 1 or Period 2 of Stage 2 PK Phase.
Arm/Group | Stage 2: Niraparib Tablet | Stage 2: Niraparib Capsule
Number analyzed (Participants) | 107 | 107
Hours*nanogram per milliliter | 17070 (57.1) | 17730 (54.1)
Statistical Analysis 1: Comparison: Stage 2: Niraparib Tablet vs Stage 2: Niraparib Capsule; Test type: Equivalence — Bioequivalence was concluded if the 90% confidence interval of the ratio of geometric least-squares means of the test (tablet) to reference (capsule) product was within 0.80 - 1.25% for AUC0-t; Ratio of geometric least square mean = 0.9594, 90% CI 2-sided [0.9199 to 1.0006] — Analysis was performed using linear mixed model with fixed effects of treatment, period, sequence, and random effect for participant nested within sequence. Ratio of geometric least square mean of niraparib tablet to niraparib capsule is presented

9. Primary Outcome: AUC(0 to Inf) for Niraparib-Stage 2 PK Phase
Description: as for outcome 2
Time Frame: Pre-dose, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose in each treatment period
Population: BE Evaluable Population. Only those participants with estimable PK parameter data available in both Periods were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Stage 2: Niraparib Tablet | Stage 2: Niraparib Capsule
Number analyzed (Participants) | 98 | 98
Hours*nanogram per milliliter | 17760 (55.3) | 18470 (53.5)
Statistical Analysis 1: Comparison: Stage 2: Niraparib Tablet vs Stage 2: Niraparib Capsule; Test type: Equivalence — Bioequivalence was concluded if the 90% confidence interval of the ratio of geometric least-squares means of the test (tablet) to reference (capsule) product was within 0.80 - 1.25% for AUC0-inf; Ratio of geometric least square mean = 0.9566, 90% CI 2-sided [0.9164 to 0.9986] — [estimate comment as in outcome 8, analysis 1]

10. Primary Outcome: Cmax for Niraparib-Stage 2 PK Phase
Description: as for outcome 3
Time Frame: Pre-dose, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose in each treatment period
Population: BE Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Stage 2: Niraparib Tablet | Stage 2: Niraparib Capsule
Number analyzed (Participants) | 108 | 108
Nanograms per milliliter | 519.5 (49.5) | 538.4 (49.4)
Statistical Analysis 1: Comparison: Stage 2: Niraparib Tablet vs Stage 2: Niraparib Capsule; Test type: Equivalence — Bioequivalence was concluded if the 90% confidence interval of the ratio of geometric least-squares means of the test (tablet) to reference (capsule) product was within 0.80 - 1.25% for Cmax; Ratio of geometric least square mean = 0.9619, 90% CI 2-sided [0.9124 to 1.0140] — [estimate comment as in outcome 8, analysis 1]

11. Primary Outcome: Tmax for Niraparib-Stage 2 PK Phase
Description: as for outcome 4
Time Frame: Pre-dose, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose in each treatment period
Population: BE Evaluable Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Stage 2: Niraparib Tablet | Stage 2: Niraparib Capsule
Number analyzed (Participants) | 108 | 108
Hours | 5.00 [1.55 to 8.00] | 4.97 [0.970 to 23.8]

12. Primary Outcome: T1/2 for Niraparib-Stage 2 PK Phase
Description: as for outcome 5
Time Frame: Pre-dose, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose in each treatment period
Population: BE Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Stage 2: Niraparib Tablet | Stage 2: Niraparib Capsule
Number analyzed (Participants) | 108 | 108
Hours | 47.94 (26.4) | 50.17 (26.1)

13. Primary Outcome: CL/F for Niraparib-Stage 2 PK Phase
Description: as for outcome 6
Time Frame: Pre-dose, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose in each treatment period
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Stage 2: Niraparib Tablet | Stage 2: Niraparib Capsule
Number analyzed (Participants) | 98 | 98
Liters per hour | 16.89 (55.3) | 16.25 (53.5)

14. Primary Outcome: Vz/F for Niraparib-Stage 2 PK Phase
Description: as for outcome 7
Time Frame: Pre-dose, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose in each treatment period
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Stage 2: Niraparib Tablet | Stage 2: Niraparib Capsule
Number analyzed (Participants) | 98 | 98
Liters | 1128 (51.1) | 1128 (50.9)

15. Primary Outcome: AUC(0-t) for Niraparib-Stage 3 PK Phase
Description: as for outcome 1
Time Frame: Pre-dose, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose in each treatment period
Population: Food Effect (FE) Evaluable Population included all participants who completed both PK periods and had sufficient PK sample collection to accurately estimate PK parameters in both periods. Participants meeting non-evaluability criteria or having significant niraparib carryover (Baseline concentration >5% of Cmax) were completely excluded from the FE Population. Only those participants with estimable PK parameter data available in both Periods were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Groups:
- Stage 3: Niraparib Tablet Fasted: Participants received a single oral dose of 300 mg niraparib tablet in a fasted state in either Period 1 or Period 2 of Stage 3 PK Phase.
- Stage 3: Niraparib Tablet Fed: Participants received a single oral dose of 300 mg niraparib tablet in a fed state with a high fat meal in either Period 1 or Period 2 of Stage 3 PK Phase.
Arm/Group | Stage 3: Niraparib Tablet Fasted | Stage 3: Niraparib Tablet Fed
Number analyzed (Participants) | 16 | 16
Hours*nanogram per milliliter | 20100 (63.9) | 25990 (52.4)
Statistical Analysis 1: Comparison: Stage 3: Niraparib Tablet Fasted vs Stage 3: Niraparib Tablet Fed; Test type: Other; Ratio of geometric least square mean = 1.3154, 90% CI 2-sided [1.1742 to 1.4735] — Analysis was performed using linear mixed model with fixed effects of treatment, period, sequence, and random effect for participant nested within sequence

16. Primary Outcome: AUC(0 to Inf) for Niraparib-Stage 3 PK Phase
Description: as for outcome 2
Time Frame: Pre-dose, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose in each treatment period
Population: FE Evaluable Population. Only those participants with estimable PK parameter data available in both Periods were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Stage 3: Niraparib Tablet Fasted | Stage 3: Niraparib Tablet Fed
Number analyzed (Participants) | 18 | 18
Hours*nanogram per milliliter | 23600 (78.5) | 29770 (65.2)
Statistical Analysis 1: Comparison: Stage 3: Niraparib Tablet Fasted vs Stage 3: Niraparib Tablet Fed; Test type: Other; Ratio of geometric least square mean = 1.2771, 90% CI 2-sided [1.1537 to 1.4137] — [estimate comment as in outcome 15, analysis 1]

17. Primary Outcome: Cmax for Niraparib-Stage 3 PK Phase
Description: as for outcome 3
Time Frame: Pre-dose, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose in each treatment period
Population: FE Evaluable Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Stage 3: Niraparib Tablet Fasted | Stage 3: Niraparib Tablet Fed
Number analyzed (Participants) | 19 | 19
Nanograms per milliliter | 704.1 (57.0) | 774.6 (47.2)
Statistical Analysis 1: Comparison: Stage 3: Niraparib Tablet Fasted vs Stage 3: Niraparib Tablet Fed; Test type: Other; Ratio of geometric least square mean = 1.1129, 90% CI 2-sided [0.9408 to 1.3164] — [estimate comment as in outcome 15, analysis 1]

18. Primary Outcome: Tmax for Niraparib-Stage 3 PK Phase
Description: as for outcome 4
Time Frame: Pre-dose, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose in each treatment period
Population: FE Evaluable Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Stage 3: Niraparib Tablet Fasted | Stage 3: Niraparib Tablet Fed
Number analyzed (Participants) | 19 | 19
Hours | 4.88 [2.97 to 7.10] | 5.97 [0.980 to 11.1]

19. Primary Outcome: T1/2 for Niraparib-Stage 3 PK Phase
Description: as for outcome 5
Time Frame: Pre-dose, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose in each treatment period
Population: FE Evaluable Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Stage 3: Niraparib Tablet Fasted | Stage 3: Niraparib Tablet Fed
Number analyzed (Participants) | 19 | 19
Hours | 46.39 (20.5) | 46.08 (22.4)

20. Primary Outcome: CL/F for Niraparib-Stage 3 PK Phase
Description: as for outcome 6
Time Frame: Pre-dose, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose in each treatment period
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Stage 3: Niraparib Tablet Fasted | Stage 3: Niraparib Tablet Fed
Number analyzed (Participants) | 18 | 18
Liters per hour | 12.71 (78.5) | 10.08 (65.2)

21. Primary Outcome: Vz/F for Niraparib-Stage 3 PK Phase
Description: as for outcome 7
Time Frame: Pre-dose, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose in each treatment period
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Stage 3: Niraparib Tablet Fasted | Stage 3: Niraparib Tablet Fed
Number analyzed (Participants) | 18 | 18
Liters | 833.8 (83.5) | 651.4 (54.3)

22. Primary Outcome: Time From Administration of the Dose to the First Quantifiable Concentration (Tlag) for Niraparib-Stage 3 PK Phase
Description: Blood samples were collected at indicated time points for pharmacokinetic assessment of tlag. Pharmacokinetic parameters were calculated using standard non-compartmental analysis.
Time Frame: Pre-dose, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose in each treatment period
Population: FE Evaluable Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Stage 3: Niraparib Tablet Fasted | Stage 3: Niraparib Tablet Fed
Number analyzed (Participants) | 19 | 19
Hours | 0.00 [0.00 to 0.970] | 0.00 [0.00 to 2.93]

23. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs-Stage 1 PK Phase (Periods 1 and 2 Only)
Description: An adverse event is any untoward medical occurrence in a clinical investigation participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. A serious adverse event (SAE) is any untoward medical occurrence that, at any dose; results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or is an important medical event. TEAE is any event that was not present prior to the initiation of study treatment or any event already present that worsens in either intensity or frequency following exposure to study treatment. TEAEs reported under Niraparib tablet and Niraparib capsule arms include TEAEs with onset date during the corresponding period (Period 1 or Period 2) in which the participant received niraparib tablet and capsule, respectively.
Time Frame: Up to 16 days
Population: Safety Population comprised of all participants who received any amount of niraparib during the Stage 1 PK Phase of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Niraparib Tablet | Stage 1: Niraparib Capsule
Number analyzed (Participants) | 29 | 29
Participants
  TEAE | 9 | 12
  Serious TEAE | 0 | 0

24. Secondary Outcome: Number of Participants With TEAEs Leading to Discontinuation -Stage 1 PK Phase (Periods 1 and 2 Only)
Description: An adverse event is any untoward medical occurrence in a clinical investigation participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. TEAE is any event that was not present prior to the initiation of study treatment or any event already present that worsens in either intensity or frequency following exposure to study treatment. Number of participants with TEAEs leading to discontinuation is reported. TEAEs reported under Niraparib tablet and Niraparib capsule arms include TEAEs with onset date during the corresponding period (Period 1 or Period 2) in which the participant received niraparib tablet and capsule, respectively.
Time Frame: Up to 16 days
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Niraparib Tablet | Stage 1: Niraparib Capsule
Number analyzed (Participants) | 29 | 29
Participants | 0 | 0

25. Secondary Outcome: Number of Participants With TEAEs and Serious TEAEs-Stage 2 PK Phase (Periods 1 and 2 Only)
Description: An adverse event is any untoward medical occurrence in a clinical investigation participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that, at any dose; results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or is an important medical event. TEAE is any event that was not present prior to the initiation of study treatment or any event already present that worsens in either intensity or frequency following exposure to study treatment. TEAEs reported under Niraparib tablet and Niraparib capsule arms include TEAEs with onset date during the corresponding period (Period 1 or Period 2) in which the participant received niraparib tablet and capsule, respectively.
Time Frame: Up to 24 days
Population: Safety Population comprised of all participants who received any amount of niraparib during the Stage 2 PK Phase of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: Niraparib Tablet | Stage 2: Niraparib Capsule
Number analyzed (Participants) | 156 | 152
Participants
  TEAE | 86 | 73
  Serious TEAE | 10 | 10

26. Secondary Outcome: Number of Participants With TEAEs-leading to Discontinuation Stage 2 PK Phase (Periods 1 and 2 Only)
Description: An adverse event is any untoward medical occurrence in a clinical investigation participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. Number of participants with TEAEs leading to discontinuation is reported. TEAEs reported under Niraparib tablet and Niraparib capsule arms include TEAEs with onset date during the corresponding period (Period 1 or Period 2) in which the participant received niraparib tablet and capsule, respectively.
Time Frame: Up to 24 days
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: Niraparib Tablet | Stage 2: Niraparib Capsule
Number analyzed (Participants) | 156 | 152
Participants | 2 | 2

27. Secondary Outcome: Number of Participants With TEAEs and Serious TEAEs-Stage 3 PK Phase (Periods 1 and 2 Only)
Description: An adverse event is any untoward medical occurrence in a clinical investigation participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that, at any dose; results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or is an important medical event. TEAE is any event that was not present prior to the initiation of study treatment or any event already present that worsens in either intensity or frequency following exposure to study treatment. TEAEs reported under Niraparib tablets under fasted and fed arms include TEAEs with onset date during the corresponding period (Period 1 or Period 2) in which the participant received niraparib tablet fasted and fed, respectively.
Time Frame: Up to 45 days
Population: Safety Population comprised of all participants who received any amount of niraparib during the Stage 3 PK Phase of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 3: Niraparib Tablet Fasted | Stage 3: Niraparib Tablet Fed
Number analyzed (Participants) | 26 | 25
Participants
  TEAE | 8 | 12
  Serious TEAE | 4 | 2

28. Secondary Outcome: Number of Participants With TEAEs-leading to Discontinuation Stage 3 PK Phase (Periods 1 and 2 Only)
Description: An adverse event is any untoward medical occurrence in a clinical investigation participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. Number of participants with TEAEs leading to discontinuation is reported. TEAEs reported under Niraparib tablets under fasted and fed arms include TEAEs with onset date during the corresponding period (Period 1 or Period 2) in which the participant received niraparib tablet fasted and fed, respectively.
Time Frame: Up to 45 days
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 3: Niraparib Tablet Fasted | Stage 3: Niraparib Tablet Fed
Number analyzed (Participants) | 26 | 25
Participants | 1 | 1

29. Secondary Outcome: Number of Participants With TEAEs and Serious TEAEs - Extension Phase
Description: An adverse event is any untoward medical occurrence in a clinical investigation participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that, at any dose; results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or is an important medical event. TEAE is any event that was not present prior to the initiation of study treatment or any event already present that worsens in either intensity or frequency following exposure to study treatment. A summary of number of participants with any TEAEs and serious TEAEs is presented. Serious TEAEs are subset of TEAEs. TEAEs were coded using the Medical Dictionary for Regulatory Affairs (MedDRA dictionary).
Time Frame: Up to approximately 5 years 5 months
Population: Safety Population comprised of all participants who received any amount of niraparib in the Open-Label Extension Phase of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Extension Phase: Niraparib Tablet | Extension Phase: Niraparib Capsule
Number analyzed (Participants) | 124 | 66
Participants
  TEAEs | 120 | 65
  Serious TEAEs | 40 | 20

30. Secondary Outcome: Number of Participants With TEAEs-leading to Discontinuation - Extension Phase
Description: An adverse event is any untoward medical occurrence in a clinical investigation participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. TEAE is any event that was not present prior to the initiation of study treatment or any event already present that worsens in either intensity or frequency following exposure to study treatment. A summary of number of participants who discontinued due to any TEAEs is presented. TEAEs were coded using the Medical Dictionary for Regulatory Affairs (MedDRA dictionary).
Time Frame: Up to approximately 5 years 5 months
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Extension Phase: Niraparib Tablet | Extension Phase: Niraparib Capsule
Number analyzed (Participants) | 124 | 66
Participants | 8 | 9

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious TEAEs and serious TEAEs were collected up to approximately 5 years 6 months.
Description: Safety Population comprised of all participants who received any amount of niraparib during the PK Phase and Extension Phase of the study. MedDRA version (v) used for PK Phase was 24.1 and Extension Phase was 26.0.
Arm/Group | Stage 1: Niraparib Tablet | Stage 1: Niraparib Capsule | Stage 2: Niraparib Tablet | Stage 2: Niraparib Capsule | Stage 3: Niraparib Tablet Fasted | Stage 3: Niraparib Tablet Fed | Extension Phase: Niraparib Tablet | Extension Phase: Niraparib Capsule
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29 | 2/156 | 5/152 | 2/26 | 0/25 | 15/124 | 3/66
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 10/156 | 10/152 | 4/26 | 2/25 | 40/124 | 20/66
Other Adverse Events (participants affected / at risk) | 2/29 | 7/29 | 49/156 | 37/152 | 6/26 | 5/25 | 113/124 | 64/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: Niraparib Tablet (N=29) | Stage 1: Niraparib Capsule (N=29) | Stage 2: Niraparib Tablet (N=156) | Stage 2: Niraparib Capsule (N=152) | Stage 3: Niraparib Tablet Fasted (N=26) | Stage 3: Niraparib Tablet Fed (N=25) | Extension Phase: Niraparib Tablet (N=124) | Extension Phase: Niraparib Capsule (N=66)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 3 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 2
Biliary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 9 | 8 | 0 | 2 | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Unresponsive to stimuli (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial necrosis marker increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: Niraparib Tablet (N=29) | Stage 1: Niraparib Capsule (N=29) | Stage 2: Niraparib Tablet (N=156) | Stage 2: Niraparib Capsule (N=152) | Stage 3: Niraparib Tablet Fasted (N=26) | Stage 3: Niraparib Tablet Fed (N=25) | Extension Phase: Niraparib Tablet (N=124) | Extension Phase: Niraparib Capsule (N=66)
Nausea (Gastrointestinal disorders) | 1 | 5 | 17 | 13 | 2 | 2 | 47 | 28
Vomiting (Gastrointestinal disorders) | 1 | 2 | 10 | 8 | 2 | 1 | 39 | 19
Fatigue (General disorders) | 1 | 2 | 12 | 8 | 0 | 0 | 34 | 22
Constipation (Gastrointestinal disorders) | 0 | 0 | 16 | 10 | 2 | 0 | 31 | 11
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 9 | 8 | 0 | 2 | 35 | 20
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 12 | 12
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 19 | 8
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 7 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 8
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 4
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 7
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 3
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 5
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 28 | 6
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 12
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 8
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 6
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT03329001/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/01/NCT03329001/SAP_002.pdf